CLINICAL TRIAL: NCT06408870
Title: Bioequivalence of the BI 1015550 Low Dose Formulation C2 and the BI 1015550 Low Dose Formulation C1 (Phase 3 Formulation) Following Oral Administration in Healthy Subjects (an Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare How 2 Different Low Dose Formulations of BI 1015550 Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0051; 2023-509951-15-00 (Registry Identifier: CTIS); U1111-1301-0913 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1015550 Formulation C1 (Reference, R) then BI 1015550 Formulation C2 (Test, T) (Experimental): For this two period crossover study arm, participants received treatment in the following order:
  Participants received a single oral dose of nerandomilast (BI 1015550), a low dose film coated tablet (formulation C1, titanium dioxide [TiO2]-containing phase III formulation, reference (R)) with 240 mL water after an overnight fast of at least 10 h (period 1).
  Participants received a single oral dose of nerandomilast (BI 10105550), a low dose film coated tablet (formulation C2, titanium dioxide [TiO2] free, test (T)) with 240 mL water after an overnight fast of at least 10 h (period 2).
  In between the treatment periods, participants went through a washout period of 10 days.
  Interventions: Drug: BI 1015550
- BI 1015550 Formulation C2 (Test, T) then BI 1015550 Formulation C1 (Reference, R) (Experimental): For this two period crossover study arm, participants received treatment in the following order:
  Participants received a single oral dose of nerandomilast (BI 10105550), a low dose film coated tablet (formulation C2, titanium dioxide [TiO2] free, test (T)) with 240 mL water after an overnight fast of at least 10 h (period 1).
  Participants received a single oral dose of nerandomilast (BI 1015550), a low dose film coated tablet (formulation C1, titanium dioxide [TiO2]-containing phase III formulation, reference (R)) with 240 mL water after an overnight fast of at least 10 h (period 2).
  In between the treatment periods, participants went through a washout period of 10 days.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — Participants received two formulations of nerandomilast separated by a washout period
  Other Names: Nerandomilast

SUMMARY:
The main objective of this trial is to establish the bioequivalence of the BI 1015550 Formulation C2 (Test, T) and the BI 1015550 Formulation C1 (Reference, R) following a single oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Female subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 7 days after last administration

Highly effective methods of contraception include:

* Use of oral hormonal contraception that prevents ovulation, plus condom
* Use of combined (estrogen and progestogen-containing) hormonal contraception that prevents ovulation (intravaginal or transdermal)
* Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants)
* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
* Sexually abstinent is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* Bilateral tubal occlusion

  - Women not of childbearing potential (WNOCBP) include:
* Permanently surgically sterilised (including hysterectomy, bilateral oophorectomy and bilateral salpingectomy)
* Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory) WNOCBP are not required to use any methods of contraception. For in vitro fertilization (IVF) and in foreign countries, female subjects should not participate in egg donation and male subjects should not participate in sperm donation from the first study drug administration, for the duration of the study and for at least 7 days after the last study drug administration.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm) at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) at screening
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to depression and suicidal behaviour
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The open-label, randomised, single-dose, two-way crossover study aimed to assess the bioequivalence of the BI 1015550 low dose Formulation C2 and the BI 1015550 low dose Formulation C1 (Phase 3 formulation) following oral administration in healthy subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment period 1
Arm/Group | BI 1015550 Formulation C1 (Reference, R) then BI 1015550 Formulation C2 (Test, T) | BI 1015550 Formulation C2 (Test, T) then BI 1015550 Formulation C1 (Reference, R)
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0
Period: Washout period
Arm/Group | BI 1015550 Formulation C1 (Reference, R) then BI 1015550 Formulation C2 (Test, T) | BI 1015550 Formulation C2 (Test, T) then BI 1015550 Formulation C1 (Reference, R)
Started | 32 | 32
Completed | 29 | 32
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 0
Period: Treatment period 2
Arm/Group | BI 1015550 Formulation C1 (Reference, R) then BI 1015550 Formulation C2 (Test, T) | BI 1015550 Formulation C2 (Test, T) then BI 1015550 Formulation C1 (Reference, R)
Started | 29 | 32
Completed | 29 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treated set was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 Formulation C1 (Reference, R) Then BI 1015550 Formulation C2 (Test, T) | BI 1015550 Formulation C2 (Test, T) Then BI 1015550 Formulation C1 (Reference, R) | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (8.1) | 35.5 (8.8) | 34.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 26 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 31 | 60
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented.
  The statistical model applied was an analysis of variance (ANOVA), with 'subjects within sequence' as a random effect and 'sequence,' 'period,' and 'treatment' as fixed effects.
Time Frame: Within 3 hours (hrs) prior to and at 15minutes (min), 30min, 45min, 1hrs, 1:15hrs, 1:30hrs, 1:45hrs, 2hrs, 2:30hrs, 3hrs, 3:30hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs, 34hrs, 48hrs, 58hrs, 72hrs, 96hrs, 120hrs, and 144hrs after nerandomilast intake.
Population: Pharmacokinetic parameter analysis set (PKS): included all subjects in the treated set (TS) who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment.
  Participants in both arms are not mutually exclusive.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/Liter (hrs*nmol/L)
Groups:
- BI 1015550 Formulation C1 (Reference, R): Participants received a single oral dose of nerandomilast (BI 1015550), a low dose film coated tablet (formulation C1, titanium dioxide [TiO2]-containing phase III formulation, reference (R)) with 240 mL water after an overnight fast of at least 10 h.
- BI 1015550 Formulation C2 (Test, T): Participants received a single oral dose of nerandomilast (BI 10105550), a low dose film coated tablet (formulation C2, titanium dioxide [TiO2] free, test (T)) with 240 mL water after an overnight fast of at least 10 h.
Arm/Group | BI 1015550 Formulation C1 (Reference, R) | BI 1015550 Formulation C2 (Test, T)
Number analyzed (Participants) | 64 | 61
hours*nanomole/Liter (hrs*nmol/L) | 1270.92 (na) — Adjusted geometric standard error = 1.04 | 1320.24 (na) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: BI 1015550 Formulation C1 (Reference, R) vs BI 1015550 Formulation C2 (Test, T); The statistical model applied was an analysis of variance (ANOVA), with 'subjects within sequence' as a random effect and 'sequence,' 'period,' and 'treatment' as fixed effects; Test type: Other; Ratio of adjusted geometric means [%] = 103.88, 90% CI 2-sided [101.08 to 106.75] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual pair geometric coefficient of variation (gCV) [%] = 9.0

2. Primary Outcome: Maximum Measured Concentration of Nerandomilast in Plasma (Cmax)
Description: Maximum measured concentration of nerandomilast in plasma (Cmax) is presented. The statistical model applied was an analysis of variance (ANOVA), with 'subjects within sequence' as a random effect and 'sequence,' 'period,' and 'treatment' as fixed effects.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1015550 Formulation C1 (Reference, R) | BI 1015550 Formulation C2 (Test, T)
Number analyzed (Participants) | 64 | 61
nanomole/Liter (nmol/L) | 218.84 (na) — Adjusted geometric standard error = 1.04 | 230.48 (na) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: BI 1015550 Formulation C1 (Reference, R) vs BI 1015550 Formulation C2 (Test, T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 105.32, 90% CI 2-sided [100.83 to 110.01] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual pair geometric coefficient of variation (gCV) [%] = 14.5

3. Secondary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented.
  The statistical model applied was an analysis of variance (ANOVA), with 'subjects within sequence' as a random effect and 'sequence,' 'period,' and 'treatment' as fixed effects.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/Liter (hrs*nmol/L)
Groups:
- BI 1015550 Formulation C2 (Test, T): Participants received a single oral dose of nerandomilast (BI 1015550), a low dose film coated tablet (formulation C2, titanium dioxide [TiO2] free, test (T)) with 240 mL water after an overnight fast of at least 10 h.
Arm/Group | BI 1015550 Formulation C1 (Reference, R) | BI 1015550 Formulation C2 (Test, T)
Number analyzed (Participants) | 64 | 61
hours*nanomole/Liter (hrs*nmol/L) | 1284.94 (na) — Adjusted geometric standard error = 1.04 | 1333.23 (na) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: BI 1015550 Formulation C1 (Reference, R) vs BI 1015550 Formulation C2 (Test, T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 103.76, 90% CI 2-sided [100.95 to 106.65] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual pair geometric coefficient of variation (gCV) [%] = 9.1

ADVERSE EVENTS:
Time Frame: For all adverse events (AEs): From first nerandomilast intake until end of residual effect period (REP), up to 7 days. For all-cause mortality: From first nerandomilast intake until end of follow-up, up to 28 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treated set was used for safety analyses.
  Participants in both arms are not mutually exclusive.
Arm/Group | BI 1015550 Formulation C1 (Reference, R) | BI 1015550 Formulation C2 (Test, T)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/61
Other Adverse Events (participants affected / at risk) | 15/64 | 10/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 Formulation C1 (Reference, R) (N=64) | BI 1015550 Formulation C2 (Test, T) (N=61)
Fatigue (General disorders) | 4 | 0
Headache (Nervous system disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT06408870/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT06408870/SAP_001.pdf